CLINICAL TRIAL: NCT02984332
Title: Short-term Muscle Disuse Induces a Rapid and Sustained Decline in Daily Myofibrillar Protein Synthesis Rates
Brief Title: Timecourse of Immobilization Experiment
Acronym: TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 650061958
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lower limb immobilisation (Experimental): All participants will undergo 7 days of unilateral leg immobilization. Participants will wear a leg brace (Donjoy X-ACT, DJO Global, USA) on one of their legs which will fix the leg at 40 degrees of flexion for the 7 days. Participants will not be allowed to remove the brace at any stage and are prohibited from bearing weight on the immobilized leg, and will ambulate on crutches throughout the week of immobilization.
  Interventions: Other: Lower limb immobilisation (leg brace)

INTERVENTIONS:
Other: Lower limb immobilisation (leg brace)

SUMMARY:
The effect of unilateral lower limb immobilisation over one week on muscle atrophy

DETAILED DESCRIPTION:
This study aims to assess the effect of one week of unilateral leg immobilization on quadriceps muscle volume and muscle protein synthesis rates. Participants wore a leg brace on one leg and ambulated on crutches during the immobilization period. Thirteen healthy young males were recruited to undertake this study.

It is currently understood that unilateral leg immobilization will result in a reduction in muscle size (Berg et al., 1996, Wall et al., 2015) and muscle protein synthesis rates after a period of disuse (de Boer et al., 2015, Glover et al., 2008). Recent research in this area has shown that even short term periods of leg immobilization (i.e. <1 week) will result in reductions in muscle size and muscle protein synthesis rates after the period of disuse (Wall et al., 2015). However we currently do not have detailed information on how muscle disuse affects muscle size and muscle protein synthesis over time during short term disuse (e.g. the first week).

The stable isotope tracer deuterium oxide (D2O) will be applied to assess cumulative muscle protein synthesis between days 0-2, 2-7 and 0-7 of the immobilization period in both the immobilized and non immobilized legs. This will be in-conjunction with bilateral vastus lateralis muscle biopsies before and after 2 and 7 days of immobilization. Furthremore, quadriceps muscle volume was assessed via MRI scans that again occured before and after 2 and 7 days of immobilization. To gain a mechanistic insight on the molecular changes during disuse a custom designed 48 well Taqman low density microarray genecard was applied to assess the transcriptional response on genes involved in muscle protein synthesis and breakdown.

ELIGIBILITY:
Inclusion Criteria:

BMI >18 and <28 no prescription medications or current illness -

Exclusion Criteria:

BMI <18 and >28 current prescription medication no history of leg injury

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Muscle size | Days 0, 2 and 7
  Quadriceps muscle volume measured via MRI

SECONDARY OUTCOMES:
Muscle protein synthesis | days 0-2, 2-7 and 0-7
  The stable isotope tracer deuterium oxide will be used to assess muscle protein synthesis. In conjunction with bilateral vastus lateralis muscle biopsies before and after 2 and 7 days which allow for the calculation of muscle protein synthesis (fractional synthesis rate) between days 0-2, 2-7 and 0-7.
Muscle strength | Pre and post immobilization
  Skeletal muscle one repetition maximum strength was assessed using standard gym equipment

CONTACTS AND LOCATIONS:
Locations (1):
- Sport & Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No